CLINICAL TRIAL: NCT06723613
Title: Effect of Exercise Program to Increase Breast Milk on Breastfeeding Self-efficacy, Breastfeeding Success and Breast Milk Quantity: A Randomized Controlled Trial
Brief Title: Exercise Program to Increase Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Principal Investigator Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/1172
Record Dates: First submitted 2024-12-01; First posted 2024-12-09 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Maternal Behavior; Breastfeeding, Exclusive; Breast Milk Expression
Keywords: Breastfeeding Self-Efficacy Scale; Breastfeeding problems; Breast Milk Quantity
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (No Intervention): Mothers in the control group will not exercise and will receive routine breastfeeding counseling.
  In the 8th and 14th weeks after birth, mothers will be subjected to; Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), LATCH- Breastfeeding Charting system, IMDAT: a tool for assessing the level of maternal milk intake scales.
- Intervention Group (Experimental): Primiparous mothers assigned to the exercise group will attend classes in groups of 8-10. Mothers will be given 1 hour (120 minutes) of exercises to increase breast milk three times a week for 6 weeks. The total training time is 18 hours. Each session will include 60 minutes of warm-up and stretching exercises and 30 minutes of relaxation exercises.
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Exercise group — Primiparous mothers assigned to the exercise group will attend classes in groups of 8-10. Mothers will be given 1 hour (120 minutes) of exercises to increase breast milk three times a week for 6 weeks. The total training time is 18 hours. Each session will include 60 minutes of warm-up and stretching exercises and 30 minutes of relaxation exercises.
  Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), LATCH-Breastfeeding Record System, IMDAT: Breast milk intake level assessment tool scales will be applied to mothers before exercise (8th week after birth) and after exercise (14th week).
  Arms: Intervention Group

SUMMARY:
In this study, the effects of an exercise program aimed at increasing breast milk on breastfeeding self-efficacy, breastfeeding success, and breast milk quantity will be evaluated.

DETAILED DESCRIPTION:
The research is a randomized controlled trial. The research will be conducted with 122 mothers who are in their 8th week postpartum and have healthy babies. Mothers in the exercise group will be given 1 hour (60 minutes) of exercise to increase breast milk three times a week for 6 weeks. The control group will be given routine breastfeeding education. Data will be collected using a sociodemographic form, Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), LATCH- Breastfeeding Charting system, IMDAT: a tool for assessing the level of maternal milk intake scale.

ELIGIBILITY:
Inclusion Criteria:

* Those who are over 18 years old,
* Who gave birth at term pregnancy (38-42 weeks),
* Who have a healthy baby,
* Who are between 8 weeks postpartum.

Exclusion Criteria:

* Those with diagnosed mental illness (e.g., antidepressants, antianxiety or antipsychotic medications),
* Those with chronic systemic illnesses,
* Those with physical illnesses that may prevent them from exercising,
* Those with any postpartum complications (hemorrhage, postpartum infection, mastitis, thromboembolic disease or postpartum psychiatric disorder).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of mothers' sociodemographic characteristics with survey before intervention | 3 months
  Mothers' sociodemographic characteristics will be collected through surveys and compared and reported
Comparison of mothers' Breastfeeding Self-Efficacy Scale averages by groups | 3 months
  Breastfeeding Self-Efficacy Scale will be applied to mothers. Breastfeeding Self-Efficacy Scale is 14-70 points (min-max) and as the score increases, it shows that mothers' breastfeeding self-sufficiency increases.
Comparison of mothers' LATCH- Breastfeeding Charting system averages by groups | 3 months
  LATCH- Breastfeeding Charting system will be applied to mothers. LATCH- Breastfeeding Charting system is 0-10 points (min-max) and as the score increases, it shows that the mothers' LATCH score increases.
Comparison of mothers' IMDAT: a tool for assessing the level of maternal milk intake averages by group. | 3 months
  IMDAT will be applied to mothers. IMDAT is 0-10 points (min-max) and the higher the score, the better the intake of breast milk.

CONTACTS AND LOCATIONS:
Locations (1):
- Seyhan Çankaya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No